CLINICAL TRIAL: NCT01745094
Title: Safety and Efficacy of Mirabegron as Add-on Therapy in Patients With Overactive Bladder Treated With Solifenacin: A Postmarketing Open-label Study in Japan
Brief Title: A Study to Evaluate the Effect of Mirabegron + Solifenacin in Overactive Bladder Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 178-CL-110
Record Dates: First submitted 2012-12-06; First posted 2012-12-07 (Estimated); Results first posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2017-12

CONDITIONS: Overactive Bladder
Keywords: mirabegron; solifenacin
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — mirabegron; Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Concomitant Group (Experimental): concomitant administration of mirabegron to solifenacin treated patients
  Interventions: Drug: mirabegron; Drug: solifenacin

INTERVENTIONS:
Drug: mirabegron — oral
  Other Names: YM178; Betanis
Drug: solifenacin — oral
  Other Names: Vesicare; YM905

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of mirabegron as add-on therapy in patients with OAB treated with solifenacin.

DETAILED DESCRIPTION:
The total duration of the study was 18 weeks, comprising a 2-week screening period and a 16-week treatment period. Patients meeting the eligibility criteria for provisional enrollment received the study drug for the screening period (solifenacin) at the same dose as that before the start of the study (2.5 or 5 mg), once daily after breakfast orally for 2 weeks. After the screening period, patients meeting the eligibility criteria for formal enrollment received the study drugs for the treatment period (solifenacin 2.5 or 5 mg and mirabegron 25 mg), once daily after breakfast orally for 16 weeks. Mirabegron dose could be increased to 50 mg at week 8 visit if the patients met all of the following criteria: (1) had an inadequate response to mirabegron at the dose of 25 mg; (2) was judged by the investigator or coinvestigator to have no safety concerns; and (3) agreed to increase the dose.

ELIGIBILITY:
Inclusion Criteria:

* Female: postmenopausal OAB outpatient
* Male: OAB outpatient who did not wish to have children at all
* Patient had been treated with solifenacin at a stable dose once daily for at least 4 weeks prior to the study
* Patient had a total OAB symptom score (OABSS ) score of ≥3 points and a Question 3 score ≥2 points

Exclusion Criteria:

* Patient had a residual urine volume of ≥100 mL or a maximum flow rate <5 mL/s, or patients with benign prostatic hyperplasia, or lower urinary tract obstruction
* Patient had serious heart disease (myocardial infarction, cardiac failure, uncontrolled angina pectoris, serious arrhythmia, use of pacemaker, etc.), liver disease, kidney disease, immunological disease, lung disease, etc. or patient had malignant tumor (except for malignant tumor that has not been treated for at least 5 y before the start of the screening period with no risk of recurrence)
* Patient had received surgical therapy that may affect the urinary tract function within 24 weeks before the start of the screening period

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2013-07-23 (Actual); Study Completion 2013-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (5):
- Japan (5):
  - Chūbu
  - Hokkaido
  - Kansai
  - Kantou
  - Kyushu

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=169

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with overactive bladder (OAB) were enrolled in 29 sites in Japan.
Groups:
- Solifenacin 2.5 mg + Mirabegron 25 mg: Participants received solifenacin 2.5 mg and mirabegron 25 mg once daily after breakfast orally for 16 weeks.
- Solifenacin 2.5 mg + Mirabegron 50 mg: Participants received solifenacin 2.5 mg and mirabegron 25 mg once daily after breakfast orally for 8 weeks. In the next 8 weeks, participants continued to receive solifenacin 2.5 mg, but received an increased dose of mirabegron 50 mg.
- Solifenacin 5 mg + Mirabegron 25 mg: Participants received solifenacin 5 mg and mirabegron 25 mg once daily after breakfast orally for 16 weeks.
- Solifenacin 5 mg + Mirabegron 50 mg: Participants received solifenacin 5 mg and mirabegron 25 mg once daily after breakfast orally for 8 weeks. In the next 8 weeks, participants continued to receive solifenacin 5 mg, but received an increased dose of mirabegron 50 mg.
Period: Overall Study
Arm/Group | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Started | 35 | 37 | 58 | 93
Completed | 30 | 37 | 46 | 90
Not Completed | 5 | 0 | 12 | 3
Not completed — Not Meeting the Eligibility Criteria | 1 | 0 | 3 | 0
Not completed — Adverse Event | 0 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 2
Not completed — Protocol Violation | 1 | 0 | 3 | 1
Not completed — Need Further Examinations Due to Biopsy | 0 | 0 | 1 | 0
Not completed — Show no Stable Solifenacin Intake | 0 | 0 | 1 | 0
Not completed — Untenable Due to Recurrent Cystitis | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAF). The SAF consisted of participants who received at least 1 dose of the study drug for the treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg | Total
Number analyzed (Participants) | 35 | 37 | 58 | 93 | 223
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.6 (8.71) | 62.8 (10.27) | 66.9 (9.47) | 63.8 (10.34) | 64.7 (9.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 32 | 45 | 79 | 186
  Male | 5 | 5 | 13 | 14 | 37
Overactive Bladder Symptom Score (OABSS) [Mean (Standard Deviation); unit: Units on a Scale] — The OABSS questionnaire was a questionnaire completed by participants with 4 questions regarding their OAB symptoms. For each participant, the OABSS total score was calculated from the sum total of the score of each question. The total score ranges from 0 to 15 with higher score indicating more symptoms. The OABSS data obtained at week 0 were used as baseline. Population: Full Analysis Set (FAS). The FAS consisted of participants who received at least 1 dose of the study drug for the treatment period, and who provided evaluable patient diary data for at least 1 efficacy variable, before and after the start of the treatment period. Participants with available data are included in the analysis.
  Units on a Scale
    number analyzed (Participants) | 33 | 37 | 55 | 93 | 218
    (all) | 7.1 (2.31) | 8.5 (2.36) | 7.5 (2.67) | 8.1 (2.45) | 7.8 (2.49)
Overactive Bladder questionnaire Short Form (OAB-q SF) Score: Symptom Severity [Mean (Standard Deviation); unit: Units on a Scale] — The OAB-q SF questionnaire was a questionnaire completed by participants composed of 2 sections: Severity Symptom and the Health-related Quality of Life (HRQL). The Severity Symptom section included 6 questions. For each participant, the symptom severity score was derived as a sum of scores for Questions 1 to 6. The total score ranges from 6 to 36 with higher symptom severity score indicating greater symptom bother. OAB-q SF data obtained at week 0 visit were used as baseline. Population: FAS participants with available data are included in the analysis.
  Units on a Scale
    number analyzed (Participants) | 33 | 37 | 55 | 93 | 218
    (all) | 33.94 (20.386) | 39.37 (20.470) | 32.12 (17.701) | 31.29 (19.205) | 33.27 (19.328)
OAB-q SF Score: Total Health-Related Quality of Life (HRQOL) [Mean (Standard Deviation); unit: Units on a Scale] — The OAB-q SF questionnaire was a questionnaire completed by participants composed of 2 sections: Severity Symptom and the HRQL. The HRQL section included 13 questions. For each participant, the total HRQL score was derived as a sum of scores for Questions 7 to 19. The total score ranges from 13 to 78 with higher total HRQL score indicating greater HRQL. OAB-q SF data obtained at week 0 visit were used as baseline. Population: FAS participants with available data are included in the analysis.
  Units on a Scale
    number analyzed (Participants) | 33 | 37 | 55 | 93 | 218
    (all) | 73.71 (18.662) | 70.31 (18.873) | 75.10 (17.708) | 76.06 (19.341) | 74.49 (18.743)
Number of Micturitions per 24 Hours [Mean (Standard Deviation); unit: micturitions] — The mean number of micturitions per 24 hours was calculated by taking the sum of all marked episodes in the patient diary where the variable "urinated" was indicated, divided by the number of days on which episodes were recorded. Population: FAS participants with available data are included in the analysis.
  micturitions
    number analyzed (Participants) | 33 | 37 | 55 | 93 | 218
    (all) | 10.38 (2.128) | 11.12 (2.722) | 9.81 (1.918) | 10.15 (2.331) | 10.26 (2.302)
Number of Urgency Episodes per 24 Hours [Mean (Standard Deviation); unit: urgency episodes] — An urgency episode was defined as a complaint of a sudden, compelling desire to pass urine, which is difficult to defer. The mean number of urgency episodes per 24 hours was calculated by taking the sum of all marked episodes in the patient diary where the variable "urgency" was indicated, divided by the number of days on which episodes were recorded. Only participants who had an urgency episode at baseline was included in the analysis. Population: FAS participants with available data are included in the analysis.
  urgency episodes
    number analyzed (Participants) | 30 | 36 | 49 | 90 | 205
    (all) | 2.86 (2.433) | 4.12 (2.586) | 2.86 (1.997) | 3.63 (2.846) | 3.42 (2.586)
Number of Incontinence Episodes per 24 Hours [Mean (Standard Deviation); unit: incontinence episodes] — An incontinence episode was defined as the complaint of any involuntary leakage of urine. The mean number of incontinence episodes per 24 hours was calculated by taking the sum of all marked episodes in the patient diary where the variable "urinary incontinence'" was indicated, divided by the number of days on which episodes were recorded. Only participants who had an incontinence episode at baseline was included in the analysis. Population: FAS participants with available data are included in the analysis.
  incontinence episodes
    number analyzed (Participants) | 14 | 28 | 29 | 60 | 131
    (all) | 1.45 (1.454) | 1.54 (1.248) | 2.09 (2.121) | 1.51 (1.520) | 1.64 (1.616)
Number of Urge Incontinence Episodes per 24 Hours [Mean (Standard Deviation); unit: urge incontinence episodes] — An urge incontinence episode was defined as any episode when both urgency and incontinence occurred concurrently. The mean number of incontinence episodes per 24 hours was calculated by taking the sum of all marked episodes in the patient diary where the variable "urgency" and "urinary incontinence'" were indicated, divided by the number of days on which episodes were recorded. Only participants who had an urge incontinence episode at baseline was included in the analysis. Population: FAS participants with available data are included in the analysis.
  urge incontinence episodes
    number analyzed (Participants) | 11 | 28 | 26 | 52 | 117
    (all) | 1.42 (1.506) | 1.42 (1.243) | 1.69 (1.366) | 1.30 (1.138) | 1.43 (1.245)
Volume Voided per Micturition [Mean (Standard Deviation); unit: mL] — The mean volume per micturition was calculated by taking the sum of the urinary volumes where the volume voided was > 0 and where "urinary incontinence" was not indicated in the patient diary, divided by the number of micturitions where the volume voided was > 0 and where "urinary incontinence" was not indicated. Only participants who had volume voided was > 0 at baseline was included in the analysis. Population: FAS participants with available data are included in the analysis.
  mL
    number analyzed (Participants) | 33 | 37 | 55 | 93 | 218
    (all) | 158.627 (47.0511) | 158.633 (43.6678) | 182.362 (56.3405) | 173.658 (47.5973) | 171.029 (49.7826)
Number of Nocturia Episodes per Night [Mean (Standard Deviation); unit: nocturia episodes] — A nocturia episode was defined as waking at night 1 or more times to void. Night time was defined as the period between bedtime and the wake-up time the following day (micturitions at the same time as the wake-up time were excluded). The mean number of nocturia episodes per night was calculated by taking the sum of nocturia episodes in the patient diary where the variable "urinated" was indicated during the night time, divided by the number of nights. Only participants who had a nocturia episode at baseline was included in the analysis. Population: FAS participants with available data are included in the analysis.
  nocturia episodes
    number analyzed (Participants) | 28 | 29 | 50 | 81 | 188
    (all) | 1.79 (1.075) | 1.55 (0.783) | 1.85 (1.006) | 1.72 (1.084) | 1.74 (1.018)
Postvoid Residual (PVR) Volume [Mean (Standard Deviation); unit: mL] — Measurement of PVR volume was made using either ultrasonography or urethral catheterization, provided that the same method was used for the same participant throughout the study.
  mL | 14.95 (23.214) | 10.51 (16.066) | 13.93 (17.188) | 12.11 (20.199) | 12.76 (19.273)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs were defined as AEs observed after the first administration of the study drugs for the treatment period. The investigator assessed the severity of AEs, including abnormal clinical laboratory values, Electrocardiogram (ECG), vital signs, as follows: Mild: No disruption of normal daily activities; Moderate: Affected normal daily activities; Severe: Inability to perform daily activities. A drug-related TEAE was a TEAE with at least a possible relationship to the study drug as assessed by the investigator.
Time Frame: From first dose of study drug up to weeks 16
Population: SAF
Measure: Count of Participants; unit: Participants
Arm/Group | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 35 | 37 | 58 | 93
Participants
  Any TEAEs | 23 | 21 | 42 | 69
  Mild | 22 | 20 | 40 | 67
  Moderate | 1 | 1 | 1 | 2
  Severe | 0 | 0 | 1 | 0
  Drug-related TEAEs | 6 | 6 | 12 | 28
  Deaths | 0 | 0 | 0 | 0
  Serious TEAEs | 1 | 1 | 5 | 4
  Drug-related Serious TEAEs | 0 | 0 | 1 | 0
  TEAEs leading to permanent discontinuation (PD) | 0 | 0 | 3 | 1
  Drug-related TEAEs leading to PD | 0 | 0 | 2 | 1

2. Secondary Outcome: Change From Baseline in OABSS Total Score
Description: The OABSS questionnaire was a questionnaire completed by participants with 4 questions regarding their OAB symptoms. For each participant, the OABSS total score was calculated from the sum total of the score of each question. The total score ranges from 0 to 15 with higher score indicating more symptoms. The OABSS data obtained at week 0 were used as baseline.
Time Frame: Baseline and week 8, 16
Population: FAS participants with available data at each time point are included in the analysis. A last visit analysis (at the end of study) was performed to ensure all patients with postbaseline data were included in the analyses. Last observation carried forward (LOCF) imputation was used for the end of study analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 33 | 37 | 55 | 93
units on a scale
  Week 8: number analyzed (Participants) | 31 | 37 | 51 | 93
  Week 8 | -3.5 (2.32) | -2.1 (2.22) | -3.5 (2.52) | -2.5 (2.32)
  Week 16: number analyzed (Participants) | 30 | 37 | 46 | 90
  Week 16 | -3.5 (2.60) | -3.9 (2.70) | -3.6 (2.90) | -4.0 (2.90)
  Week 16 (LOCF): number analyzed (Participants) | 33 | 37 | 53 | 93
  Week 16 (LOCF) | -3.4 (2.95) | -3.9 (2.70) | -3.6 (2.86) | -4.0 (2.90)

3. Secondary Outcome: Number of Participants Who Achieved Normalization for OABSS Total Score
Description: Normalization for OABSS Total Score was defined as OABSS total score ≤ 2 or OABSS Question 3 score ≤ 1.
Time Frame: Week 8 and 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 33 | 37 | 55 | 93
Participants
  Week 8: number analyzed (Participants) | 31 | 37 | 51 | 93
  Week 8 | 19 | 8 | 28 | 26
  Week 16: number analyzed (Participants) | 30 | 37 | 46 | 90
  Week 16 | 18 | 16 | 27 | 48
  Week 16 (LOCF): number analyzed (Participants) | 33 | 37 | 53 | 93
  Week 16 (LOCF) | 19 | 16 | 29 | 49

4. Secondary Outcome: Change From Baseline in Overactive Bladder Questionnaire Short Form (OAB-q SF) Severity Score
Description: The OAB-q SF questionnaire was a questionnaire completed by participants composed of 2 sections: Severity Symptom and the Health-related Quality of Life (HRQL). The Severity Symptom section included 6 questions. For each participant, the symptom severity score was derived as a sum of scores for Questions 1 to 6. The total score ranges from 6 to 36 with higher symptom severity score indicating greater symptom bother. OAB-q SF data obtained at week 0 visit were used as baseline.
Time Frame: Baseline and week 8, 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 33 | 37 | 55 | 93
units on a scale
  Week 8: number analyzed (Participants) | 31 | 37 | 51 | 93
  Week 8 | -19.46 (16.735) | -12.52 (20.926) | -15.29 (14.348) | -10.39 (17.222)
  Week 16: number analyzed (Participants) | 30 | 37 | 46 | 90
  Week 16 | -21.00 (19.557) | -22.25 (20.877) | -17.68 (15.930) | -16.56 (18.171)
  Week 16 (LOCF): number analyzed (Participants) | 33 | 37 | 53 | 93
  Week 16 (LOCF) | -21.21 (18.631) | -22.25 (20.877) | -17.55 (16.253) | -16.31 (18.034)

5. Secondary Outcome: Change From Baseline in OAB-q SF Total HRQL Score
Description: The OAB-q SF questionnaire was a questionnaire completed by participants composed of 2 sections: Severity Symptom and the HRQL. The HRQL section included 13 questions. For each participant, the total HRQL score was derived as a sum of scores for Questions 7 to 19. The total score ranges from 13 to 78 with higher total HRQL score indicating greater HRQL. OAB-q SF data obtained at week 0 visit were used as baseline.
Time Frame: Baseline and week 8, 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 33 | 37 | 55 | 93
units on a scale
  Week 8: number analyzed (Participants) | 31 | 37 | 51 | 93
  Week 8 | 15.14 (12.786) | 9.31 (15.559) | 12.43 (15.449) | 6.14 (13.797)
  Week 16: number analyzed (Participants) | 30 | 37 | 46 | 90
  Week 16 | 17.54 (13.349) | 16.72 (16.439) | 14.72 (16.428) | 12.72 (17.170)
  Week 16 (LOCF): number analyzed (Participants) | 33 | 37 | 53 | 93
  Week 16 (LOCF) | 17.34 (13.005) | 16.72 (16.439) | 13.88 (16.080) | 12.56 (17.022)

6. Secondary Outcome: Change From Baseline in the Number of Micturitions Per 24 Hours
Description: Participants completed the patient diary (paper document) for 3 days immediately before each visit. The mean number of micturitions per 24 hours was calculated by taking the sum of all marked episodes in the patient diary where the variable "urinated" was indicated, divided by the number of days on which episodes were recorded.
Time Frame: Baseline and week 4, 8, 12, 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micturitions
Arm/Group | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 33 | 37 | 55 | 93
micturitions
  Week 4: number analyzed (Participants) | 31 | 37 | 53 | 93
  Week 4 | -0.34 (1.576) | -0.98 (1.977) | -1.33 (1.604) | -1.02 (1.666)
  Week 8: number analyzed (Participants) | 30 | 37 | 47 | 93
  Week 8 | -1.69 (1.690) | -1.31 (1.862) | -1.74 (1.586) | -1.32 (1.656)
  Week 12: number analyzed (Participants) | 31 | 37 | 45 | 90
  Week 12 | -1.98 (1.667) | -2.40 (1.997) | -1.50 (1.850) | -1.75 (2.136)
  Week 16: number analyzed (Participants) | 30 | 37 | 46 | 90
  Week 16 | -2.06 (1.677) | -2.36 (2.106) | -1.90 (1.920) | -2.13 (2.118)
  Week 16 (LOCF) | -1.89 (1.789) | -2.36 (2.106) | -1.94 (1.792) | -2.12 (2.094)

7. Secondary Outcome: Number for Participants Who Achieved Normalization of the Number of Micturitions Per 24 Hours
Description: Normalization for the mean number of micturitions per 24 hours was defined as < 8 micturitions per 24 hours.
Time Frame: Week 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 33 | 37 | 55 | 93
Participants | 10 | 17 | 23 | 40

8. Secondary Outcome: Change From Baseline in the Number of Urgency Episodes Per 24 Hours
Description: Participants completed the patient diary (paper document) for 3 days immediately before each visit. An urgency episode was defined as a complaint of a sudden, compelling desire to pass urine, which is difficult to defer. The mean number of urgency episodes per 24 hours was calculated by taking the sum of all marked episodes in the patient diary where the variable "urgency" was indicated, divided by the number of days on which episodes were recorded. Only participants who had an urgency episode at baseline was included in the analysis.
Time Frame: Baseline and week 4, 8, 12, 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: urgency episodes
Arm/Group | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 30 | 36 | 49 | 90
urgency episodes
  Week 4: number analyzed (Participants) | 28 | 36 | 48 | 90
  Week 4 | -1.15 (1.843) | -1.26 (1.927) | -1.45 (1.790) | -1.43 (2.057)
  Week 8: number analyzed (Participants) | 27 | 36 | 43 | 90
  Week 8 | -1.77 (0.969) | -1.49 (1.897) | -1.76 (1.490) | -1.37 (2.189)
  Week 12: number analyzed (Participants) | 28 | 36 | 41 | 87
  Week 12 | -1.95 (1.279) | -2.55 (2.162) | -1.89 (1.674) | -1.88 (2.576)
  Week 16: number analyzed (Participants) | 27 | 36 | 42 | 87
  Week 16 | -1.77 (1.253) | -2.59 (2.201) | -1.93 (1.759) | -2.06 (2.419)
  Week 16 (LOCF) | -1.57 (1.382) | -2.59 (2.201) | -1.93 (1.877) | -2.02 (2.392)

9. Secondary Outcome: Number for Participants Who Achieved Normalization of the Number of Urgency Episodes Per 24 Hours
Description: Normalization for the mean number of urgency episodes per 24 hours was defined as no urgency episode per 24 hours.
Time Frame: Week 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 33 | 37 | 55 | 93
Participants | 16 | 13 | 31 | 38

10. Secondary Outcome: Change From Baseline in the Number of Incontinence Episodes Per 24 Hours
Description: Participants completed the patient diary (paper document) for 3 days immediately before each visit. An incontinence episode was defined as the complaint of any involuntary leakage of urine. The mean number of incontinence episodes per 24 hours was calculated by taking the sum of all marked episodes in the patient diary where the variable "urinary incontinence'" was indicated, divided by the number of days on which episodes were recorded. Only participants who had an incontinence episode at baseline was included in the analysis.
Time Frame: Baseline and week 4, 8, 12, 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: incontinence episodes
Arm/Group | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 14 | 28 | 29 | 60
incontinence episodes
  Week 4: number analyzed (Participants) | 13 | 28 | 28 | 60
  Week 4 | -0.85 (0.675) | -0.55 (0.787) | -1.12 (1.141) | -0.64 (1.032)
  Week 8: number analyzed (Participants) | 12 | 28 | 23 | 60
  Week 8 | -1.06 (0.983) | -0.73 (0.842) | -1.26 (1.453) | -0.76 (1.273)
  Week 12: number analyzed (Participants) | 13 | 28 | 22 | 58
  Week 12 | -1.31 (1.236) | -1.04 (1.177) | -1.03 (1.238) | -0.93 (1.248)
  Week 16: number analyzed (Participants) | 12 | 28 | 22 | 58
  Week 16 | -1.22 (1.076) | -1.08 (1.168) | -1.32 (1.517) | -1.08 (1.068)
  Week 16 (LOCF) | -1.07 (1.064) | -1.08 (1.168) | -1.32 (1.505) | -1.06 (1.055)

11. Secondary Outcome: Number for Participants Who Achieved Normalization of the Number of Incontinence Episodes Per 24 Hours
Description: Normalization for the mean number of incontinence episodes per 24 hours was defined as no incontinence episode per 24 hours.
Time Frame: Week 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 33 | 37 | 55 | 93
Participants | 10 | 21 | 19 | 46

12. Secondary Outcome: Change From Baseline in the Number of Urge Incontinence Episodes Per 24 Hours
Description: Participants completed the patient diary (paper document) for 3 days immediately before each visit. An urge incontinence episode was defined as any episode when both urgency and incontinence occurred concurrently. The mean number of incontinence episodes per 24 hours was calculated by taking the sum of all marked episodes in the patient diary where the variable "urgency" and "urinary incontinence'" were indicated, divided by the number of days on which episodes were recorded. Only participants who had an urge incontinence episode at baseline was included in the analysis.
Time Frame: Baseline and week 4, 8, 12, 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: urge incontinence episodes
Arm/Group | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 11 | 28 | 26 | 52
urge incontinence episodes
  Week 4: number analyzed (Participants) | 10 | 28 | 25 | 52
  Week 4 | -0.87 (0.689) | -0.50 (0.756) | -0.77 (1.220) | -0.82 (1.055)
  Week 8: number analyzed (Participants) | 10 | 28 | 20 | 52
  Week 8 | -1.17 (1.045) | -0.65 (0.793) | -1.07 (1.068) | -0.72 (1.208)
  Week 12: number analyzed (Participants) | 10 | 28 | 19 | 50
  Week 12 | -1.30 (1.252) | -0.94 (1.115) | -0.84 (0.996) | -0.91 (1.160)
  Week 16: number analyzed (Participants) | 10 | 28 | 19 | 50
  Week 16 | -1.07 (0.940) | -1.00 (1.089) | -1.11 (1.089) | -0.96 (1.040)
  Week 16 (LOCF) | -0.97 (0.948) | -1.00 (1.089) | -1.04 (1.412) | -0.94 (1.027)

13. Secondary Outcome: Change From Baseline in the Volume Voided Per Micturition
Description: Participants completed the patient diary (paper document) for 3 days immediately before each visit. The mean volume per micturition was calculated by taking the sum of the urinary volumes where the volume voided was > 0 and where "urinary incontinence" was not indicated in the patient diary, divided by the number of micturitions where the volume voided was > 0 and where "urinary incontinence" was not indicated. Only participants who had volume voided was > 0 at baseline was included in the analysis.
Time Frame: Baseline and week 8, 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 33 | 37 | 55 | 93
mL
  Week 8: number analyzed (Participants) | 30 | 37 | 47 | 93
  Week 8 | 22.120 (26.2220) | 19.380 (31.5492) | 33.781 (32.6029) | 24.821 (35.8941)
  Week16: number analyzed (Participants) | 30 | 37 | 45 | 90
  Week16 | 28.532 (32.2243) | 33.031 (38.2492) | 35.780 (33.8236) | 36.921 (43.8896)
  Week 16 (LOCF): number analyzed (Participants) | 31 | 37 | 50 | 93
  Week 16 (LOCF) | 29.865 (32.5400) | 33.031 (38.2492) | 34.118 (32.6790) | 36.957 (43.6344)

14. Secondary Outcome: Change From Baseline in the Number of Nocturia Episodes Per Night
Description: Participants completed the patient diary (paper document) for 3 days immediately before each visit. A nocturia episode was defined as waking at night 1 or more times to void. Night time was defined as the period between bedtime and the wake-up time the following day (micturitions at the same time as the wake-up time were excluded). The mean number of nocturia episodes per night was calculated by taking the sum of nocturia episodes in the patient diary where the variable "urinated" was indicated during the night time, divided by the number of nights. Only participants who had a nocturia episode at baseline was included in the analysis.
Time Frame: Baseline and week 4, 8, 12, 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nocturia episodes
Groups:
- Solifenacin 2.5 mg + Mirabegron 25 mg: Patients received solifenacin 2.5 mg and mirabegron 25 mg once daily after breakfast orally for 16 weeks.
- Solifenacin 5 mg + Mirabegron 25 mg: Patients received solifenacin 5 mg and mirabegron 25 mg once daily after breakfast orally for 16 weeks.
Arm/Group | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 28 | 29 | 50 | 81
nocturia episodes
  Week 4: number analyzed (Participants) | 26 | 29 | 48 | 81
  Week 4 | 0.17 (1,122) | -0.07 (0.787) | -0.45 (0.709) | -0.27 (0.738)
  Week 8: number analyzed (Participants) | 25 | 29 | 43 | 81
  Week 8 | -0.38 (0.681) | -0.21 (0.688) | -0.37 (0.682) | -0.44 (0.825)
  Week 12: number analyzed (Participants) | 26 | 29 | 41 | 78
  Week 12 | -0.35 (0.704) | -0.48 (0.796) | -0.29 (0.829) | -0.58 (0.916)
  Week 16: number analyzed (Participants) | 25 | 29 | 42 | 78
  Week 16 | -0.38 (0.881) | -0.31 (0.674) | -0.44 (0.813) | -0.61 (0.992)
  Week 16 (LOCF) | -0.43 (0.847) | -0.31 (0.674) | -0.44 (0.812) | -0.60 (0.982)

15. Secondary Outcome: Change From Baseline in Postvoid Residual (PVR) Volume
Description: Measurement of PVR volume was made using either ultrasonography or urethral catheterization, provided that the same method was used for the same participant throughout the study.
Time Frame: Baseline and week 4, 8, 12, 16
Population: SAF
Measure: Mean (Standard Deviation); unit: mL
Groups:
- Solifenacin 5 mg + Mirabegron 50 mg: Participants received solifenacin 5 mg and mirabegron 25 mg once daily after breakfast orally for 8 weeks. In the next 8 weeks, participants continued to receive solifenacin 5 mg, but received an increased dose of mirabegron 50 mg."
Arm/Group | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
Number analyzed (Participants) | 35 | 37 | 58 | 93
mL
  Week 4: number analyzed (Participants) | 34 | 37 | 54 | 93
  Week 4 | -4.95 (18.078) | 5.88 (17.709) | 13.78 (35.702) | 4.36 (20.797)
  Week 8: number analyzed (Participants) | 31 | 37 | 51 | 93
  Week 8 | -2.83 (19.442) | 5.07 (19.512) | 11.05 (32.310) | 1.87 (13.428)
  Week 12: number analyzed (Participants) | 31 | 37 | 47 | 92
  Week 12 | -2.53 (21.047) | 5.29 (22.163) | 6.51 (22.067) | 1.17 (17.997)
  Week 16: number analyzed (Participants) | 30 | 37 | 46 | 90
  Week 16 | 0.63 (24.102) | 3.96 (14.897) | 7.31 (22.754) | 3.60 (24.223)
  Week 16 (LOCF): number analyzed (Participants) | 35 | 37 | 56 | 93
  Week 16 (LOCF) | -0.42 (23.576) | 3.96 (14.897) | 8.00 (28.833) | 3.17 (24.144)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to week 16
Description: Safety Analysis Set (SAF). The SAF consisted of participants who received at least 1 dose of the study drug for the treatment period.
Arm/Group | Solifenacin 2.5 mg + Mirabegron 25 mg | Solifenacin 2.5 mg + Mirabegron 50 mg | Solifenacin 5 mg + Mirabegron 25 mg | Solifenacin 5 mg + Mirabegron 50 mg
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/37 | 0/58 | 0/93
Serious Adverse Events (participants affected / at risk) | 1/35 | 1/37 | 5/58 | 4/93
Other Adverse Events (participants affected / at risk) | 23/35 | 21/37 | 39/58 | 67/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Solifenacin 2.5 mg + Mirabegron 25 mg (N=35) | Solifenacin 2.5 mg + Mirabegron 50 mg (N=37) | Solifenacin 5 mg + Mirabegron 25 mg (N=58) | Solifenacin 5 mg + Mirabegron 50 mg (N=93)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0
Blood urea increased (Investigations) | 0 | 0 | 1 | 0
ECG ST segment depression (Investigations) | 0 | 0 | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Solifenacin 2.5 mg + Mirabegron 25 mg (N=35) | Solifenacin 2.5 mg + Mirabegron 50 mg (N=37) | Solifenacin 5 mg + Mirabegron 25 mg (N=58) | Solifenacin 5 mg + Mirabegron 50 mg (N=93)
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 2
Dry eye (Eye disorders) | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 5 | 7
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Thirst (General disorders) | 1 | 0 | 1 | 3
Cystitis (Infections and infestations) | 3 | 1 | 1 | 4
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 3 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 3 | 3
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 1 | 3
Blood bilirubin increased (Investigations) | 0 | 1 | 2 | 0
Blood cholesterol increased (Investigations) | 2 | 2 | 0 | 3
Blood creatine phosphokinase increased (Investigations) | 4 | 5 | 6 | 13
Blood creatinine increased (Investigations) | 1 | 0 | 1 | 3
Blood potassium increased (Investigations) | 0 | 0 | 1 | 2
Blood pressure increased (Investigations) | 0 | 0 | 2 | 0
Blood urea increased (Investigations) | 3 | 3 | 8 | 15
Blood uric acid decreased (Investigations) | 0 | 1 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 3 | 3 | 3 | 8
Glucose urine present (Investigations) | 2 | 0 | 3 | 3
Platelet count increased (Investigations) | 1 | 0 | 0 | 0
Protein urine present (Investigations) | 0 | 2 | 0 | 0
Urinary sediment abnormal (Investigations) | 5 | 1 | 3 | 7
White blood cell count decreased (Investigations) | 2 | 3 | 1 | 6
White blood cell count increased (Investigations) | 1 | 0 | 1 | 0
White blood cells urine positive (Investigations) | 2 | 0 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 2 | 1
Headache (Nervous system disorders) | 0 | 1 | 1 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 4 | 3 | 5 | 6
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi center data. Sponsor must receive a site's manuscript prior to publication for review and comment.